CLINICAL TRIAL: NCT03923790
Title: Stroke Telemedicine Outpatient Program (STOP) for Blood Pressure Reduction
Brief Title: Stroke Telemedicine Outpatient Prevention Program for Blood Pressure Reduction
Acronym: STOP-Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Anjail Z Sharrief, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-18-0925
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Results first posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-10

CONDITIONS: Stroke Prevention; Blood Pressure; Telemedicine; Psychosocial Impairment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- STOP model (Experimental): Pharmacist evaluates patient prior to discharge and a nurse navigator contacts patient 72 hours after discharge. Patient receives educational packet and a blue tooth enabled BP monitor with an iPad. A video telehealth visit occurs 7 days after discharge attended by a nurse practitioner (NP) or MD , social worker (SW), and pharmacist. The NP and pharmacist review the BP data to determine the need for medication adjustment. The SW assesses the need for resources. BP is reviewed via an online portal every 2 weeks until average BP is < 130/80mmHg, then monthly. Uncontrolled BP prompts a call from the pharmacist to discuss medication adherence and titration. Subsequent video telehealth visits occur 1 month, 3 months, and 5 months after enrollment.
  Interventions: Behavioral: Educational Packet; Behavioral: Phone call at 72 hours by discharge nurse navigator; Behavioral: Telehealth visit at 7 days, 1 month, 3 months, and 5 months after discharge; Behavioral: Educational messages every other week; Diagnostic Test: BP monitoring by QardioARM with periodic transmission of BP data
- Usual Care (Active Comparator): Pharmacist evaluates patient prior to discharge and a nurse navigator contacts patient 72 hours after discharge. Patient receives educational packet.
  Interventions: Behavioral: Educational Packet; Behavioral: Phone call at 72 hours by discharge nurse navigator

INTERVENTIONS:
Behavioral: Educational Packet — The patient will receive an educational packet.
Behavioral: Phone call at 72 hours by discharge nurse navigator — Patients will receive a phone call at 72 hours by the discharge nurse navigator (standard of care) to assure that they have received their medications and follow-up appointments
Behavioral: Telehealth visit at 7 days, 1 month, 3 months, and 5 months after discharge — A stroke prevention trained nurse practitioner or MD or social worker will review the participant's hospital records and depression, dietary, and sleep apnea screens,will reinforce the care plan based on patient-specific needs.They will counsel patients on salt reduction, the Mediterranean diet, and the importance of diet and exercise for stroke prevention.Along with the pharmacist they will also review the BP data to determine the need for medication adjustment and will discuss the side effects and interactions.The social worker will assess the need for medication assistance and other resources. The care plan will be shared with primary care providers (PCP)and patients will be referred to a PCP if they do not have one. The social worker will also will assist uninsured patients in applying for Texas County Indigent Care programs.
  Arms: STOP model
Behavioral: Educational messages every other week — The messages will be sent to the participants cellular phones and will contain one of the following: a reminder to monitor BP, information from about lifestyle and diet for BP reduction, or a message from the pharmacist about medication adherence
  Arms: STOP model
Diagnostic Test: BP monitoring by QardioARM with periodic transmission of BP data — Participants will be prompted to transmit BP logs through the telemonitoring device every 2 weeks until average BP is < 130/80, then monthly thereafter. Uncontrolled BP will prompt a call from the pharmacist to discuss medication adherence and the need for further titration.
  Arms: STOP model

SUMMARY:
The purpose of this pilot trial is to compare post-stroke care blood pressure (BP) treatment using an interdisciplinary telehealth model [called the Stroke Telemedicine Outpatient Program (STOP) for Blood Pressure Reduction] to usual care in stroke patients at risk for uncontrolled BP. The intervention will address general and stroke-related factors associated with racial disparities in BP control. We will assess feasibility of implementation of the trial and will use the measures and outcomes assessed in the pilot to examine knowledge gaps.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic and hemorrhagic stroke patients
* Presence of at least one of the following high risk criteria: uninsured, Medicaid payer status, small vessel ischemic stroke, hypertensive ICH)
* Age ≥ 18; presence of hypertension (by clinical history or hospital BP ≥140/90 on two occasions)
* Plan to discharge home after stroke
* Ability to provide consent (patient or caregiver)
* Ability to communicate in English

Exclusion Criteria:

* modified Rankin scale > 4 at the time of enrollment (severe disability)
* life expectancy < 1 year or terminal illness,
* eGFR < 30 at time of discharge
* pregnancy
* symptomatic flow limiting carotid stenosis without plan for intervention
* urine toxicology positive for cocaine or methamphetamine or recent use
* long-term BP goal ≥ 130/80 mmHg according to clinical team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjail Sharrief, Principal Investigator — The University Of Texas Health Science Center of Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- STOP Model: Pharmacist evaluates patient prior to discharge and a nurse navigator contacts patient 72 hours after discharge. Patient receives educational packet and a blue tooth enabled BP monitor with an iPad and will also receive educational messages every other week by phone. A video telehealth visit occurs 7 days after discharge attended by a nurse practitioner (NP) or MD , social worker (SW), and pharmacist. The NP and pharmacist review the BP data to determine the need for medication adjustment. The SW assesses the need for resources. BP is reviewed via an online portal every 2 weeks until average BP is < 130/80mmHg, then monthly. Uncontrolled BP prompts a call from the pharmacist to discuss medication adherence and titration. Subsequent video telehealth visits occur 1 month, 3 months, and 5 months after enrollment.
Period: Overall Study
Arm/Group | STOP Model | Usual Care
Started | 42 | 41
Completed | 27 | 17
Not Completed | 15 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STOP Model | Usual Care | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 36 | 71
  >=65 years | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (11.6) | 53.4 (10.1) | 54.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 43
  Male | 22 | 18 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 9 | 20
  Not Hispanic or Latino | 31 | 31 | 62
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 20 | 17 | 37
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 6 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 41 | 83
Number of participants who are insured [Count of Participants; unit: Participants] | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Daytime Ambulatory Systolic Blood Pressure
Description: Blood pressure will be assessed with an ambulatory blood pressure monitor (ABPM).
Time Frame: 6 months after enrollment
Population: Data for this outcome measure were not collected for 16 in the STOP Model arm and 25 in the Usual Care arm.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | STOP Model | Usual Care
Number analyzed (Participants) | 26 | 16
millimeters of mercury (mmHg) | 123.6 (16.7) | 128.3 (19.7)

2. Secondary Outcome: Daytime Ambulatory Diastolic Blood Pressure
Description: Blood pressure will be assessed with an ambulatory blood pressure monitor (ABPM).
Time Frame: 6 months
Population: Data for this outcome measure were not collected for 16 in the STOP Model arm and 25 in the Usual Care arm.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | STOP Model | Usual Care
Number analyzed (Participants) | 26 | 16
millimeters of mercury (mmHg) | 75.1 (9.6) | 76.5 (13.7)

3. Secondary Outcome: Night Time Ambulatory Systolic Blood Pressure
Description: Blood pressure will be assessed with an ambulatory blood pressure monitor (ABPM).
Time Frame: 6 months
Population: Data for this outcome measure were not collected for 16 in the STOP Model arm and 29 in the Usual Care arm.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | STOP Model | Usual Care
Number analyzed (Participants) | 26 | 12
millimeters of mercury (mmHg) | 117.3 (16) | 119.3 (19.3)

4. Secondary Outcome: Nighttime Diastolic Blood Pressure
Description: Blood pressure will be assessed with an ambulatory blood pressure monitor (ABPM).
Time Frame: 6 months
Population: Data for this outcome measure were not collected for 16 in the STOP Model arm and 29 in the Usual Care arm.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | STOP Model | Usual Care
Number analyzed (Participants) | 26 | 12
millimeters of mercury (mmHg) | 69.4 (8.9) | 68 (13.7)

5. Secondary Outcome: Body Mass Index(BMI)
Description: BMI will be calculated from height and weight.
Time Frame: 6 months
Population: Data for this outcome measure were not collected for 22 in the STOP Model arm and 29 in the Usual Care arm.
Measure: Mean (Standard Deviation); unit: kilograms/meter^2 (kg/m^2)
Arm/Group | STOP Model | Usual Care
Number analyzed (Participants) | 20 | 12
kilograms/meter^2 (kg/m^2) | 33.8 (7.4) | 27.7 (3.9)

6. Secondary Outcome: Number of Participants With Recurrent Vascular Events (Stroke, Myocardial Infarction, Acute Cardiac Death)
Description: Recurrent vascular events include stroke, myocardial infarction, or acute cardiac death.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | STOP Model | Usual Care
Number analyzed (Participants) | 42 | 41
Participants | 3 | 2

7. Secondary Outcome: Number of Participants With Acute Healthcare Utilization
Description: Acute healthcare utilization includes hospital readmission and acute care visits to emergency room and/or urgent care.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | STOP Model | Usual Care
Number analyzed (Participants) | 42 | 41
Participants | 2 | 2

8. Other Pre Specified Outcome: Caregiver Burden as Assessed by the Zarit Caregiver Burden Questionnaire
Time Frame: 6 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Medication Adherence as Assessed by the Morisky Medication Adherence Scale (MMAS)
Time Frame: 6 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Self-efficacy for Taking Medication as Prescribed as Assessed by the Medication Adherence Self-Efficacy Scale (MASES)
Time Frame: 6 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Self-efficacy for Taking Medication as Prescribed as Assessed by the Medication Adherence Self-Efficacy Scale (MASES)
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: Mortality data were collected for all participants who were randomized. Serious Adverse Event data and Other (Not Including Serious) Adverse Event data were collected for participants who completed the study.
Arm/Group | STOP Model | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/42 | 0/41
Serious Adverse Events (participants affected / at risk) | 4/27 | 2/17
Other Adverse Events (participants affected / at risk) | 1/27 | 2/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STOP Model (N=27) | Usual Care (N=17)
Hospitalization (General disorders) | 2 (2) | 2 (2)
Hospitalization due to injury from fall (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STOP Model (N=27) | Usual Care (N=17)
Fall (General disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT03923790/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT03923790/ICF_000.pdf